CLINICAL TRIAL: NCT04881708
Title: Post-Surgical Based Efforts to Reduce Preventable Readmissions and Optimize Length of Stay
Acronym: RPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Janani S. Reisenauer, Assistant Professor of Surgery, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-000817
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current Care Group (No Intervention): The current care group will receive the standard of care currently in place within the subspecialty practices in the Department of Surgery, Mayo Clinic Rochester. This includes postoperative inpatient care directed by the surgical team, including timing of discharge and follow-up.
- Remote Care Group (Active Comparator): Patients randomized to the remote monitoring arm will engage in a Connected Care Remote Patient Monitoring (RPM) Complex Care program. RPM Complex Care programs utilize established and standardized equipment, logistics/reverse logistic, engagement methods, and nursing clinical practice. Use of RPM Complex Care programs in this manner, is considered standard practice. Patients will be monitored for 30 days by the Connected Care nursing team as is standard for surgical RPM Complex Care programs.
  Interventions: Device: Remote Monitoring

INTERVENTIONS:
Device: Remote Monitoring — Subjects assigned to the Remote Care group will receive education from a clinical nurse from Mayo Clinic's Department of Connected Care on use of the equipment as part of Remote Monitoring. The equipment will be shipped along with instructions and Welcome Letter describing the Mayo Clinic Remote Patient Monitoring program. The Remote Patient Monitoring kit includes a digital tablet, a blood pressure cuff, a thermometer, a pulse oximeter, and a weight scale. Subjects will be contacted by phone at the end of the study to be instructed how to return the kit by mail.
  Arms: Remote Care Group

SUMMARY:
The investigators believe that hospital readmissions for intermediate- to high-complexity surgeries can be reduced by remote patient monitoring follow-up post-discharge, which involves daily touchpoints with a clinical nurse, vital sign evaluation and a symptom directed communication escalation process.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years of age)
* Undergoing one of the following inpatient elective surgery procedures: abdominal wall reconstruction, bariatrics, hepatectomy, pancreatectomy, aortic surgery, lower extremity bypass, esophagectomy and colectomy at Mayo Clinic Rochester.
* Must be willing to actively work with RPM nurses with vital sign capturing.

Exclusion Criteria:

* Have uncontrolled mental illness and/or drug or alcohol abuse
* Reside in a long-term care facility
* Are being actively followed by dialysis or transplant services
* Pregnant
* Are being actively treated for cancer, receiving chemo or radiation therapy during the remote monitoring
* Are identified as end-of-life by provider
* Have dementia, cognitive impairment, or physical condition that limits ability to use home remote monitoring equipment independently or interact with remote patient monitoring staff (unless a caregiver commits to assisting daily).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Length of Stay | Until hospital discharge, typically 3 to 7 days
  Track the length of hospital stay in each group and compare.

SECONDARY OUTCOMES:
30-day readmission rates | 30 day
  Evaluate the number of patients that are readmitted to the hospital in each group and compare.

CONTACTS AND LOCATIONS:
Overall Officials: Janani Reisenauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials